CLINICAL TRIAL: NCT01407081
Title: SMARTease Trial - Turning SMART Goals Into Smart Actions: Evaluating Stroke Help Distance Interventions to Improve Cognitive Performance Post-Stroke
Brief Title: SMARTease Trial: Evaluating Stroke Help Distance Interventions to Improve Cognitive Performance Post-Stroke
Acronym: SMARTease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: IWK Health Centre (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Gail Eskes, Dr. Gail Eskes, Professor, Department of Psychiatry, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDHA-RS/2012-040
Record Dates: First submitted 2011-06-23; First posted 2011-08-01 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Cognitive Impairment; Stroke
Keywords: cognitive rehabilitation; SMART goals; telehealth
MeSH Terms: conditions — Cognitive Dysfunction; Stroke | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Training (Experimental): telerehabilitation cognitive strategy training
  Interventions: Behavioral: Telerehabilitation Cognitive Strategy Training

INTERVENTIONS:
Behavioral: Telerehabilitation Cognitive Strategy Training — The strategy intervention is a 16-week program during which a trained rehabilitation coach speaks by telephone to the stroke participant and their caregiver twice a week (one approximately 45-minute 'training' call and one approximately 15-minute 'update' call). Rehabilitation discussions during the training calls will follow a detailed protocol and focus each week on the stroke education and cognitive strategy training information provided in each section of the manual provided to the participants.
  Other Names: cognitive rehabilitation

SUMMARY:
The purpose of this study is to provide evidence for the feasibility and initial effectiveness of a manualized, telephone-based (telehealth) approach to the delivery of cognitive interventions (SMARTease) targeted to improve cognitive performance in daily activities after stroke.

DETAILED DESCRIPTION:
An initial brief screening interview will be completed with the potential participant by telephone to determine whether or not the individual meets the criteria for the study.

In an initial onsite visit, informed consent will be obtained from both the stroke survivor and their study partner and baseline evaluations will be completed with the stroke survivor, including a baseline cognitive assessment and setting goals to work on during the study period. Then the introductory section of the study Handbook (Making the Most of Your Memory) which includes procedural information on the Stroke Help Program will be reviewed with the stroke survivor and study partner. A study Handbook and a large button speaker phone will be provided to the stroke survivor/partner pair to ensure that both members of the participant-caregiver team can listen to the rehabilitation coach without having to be concerned with holding a handset (an action that may be difficult for some stroke survivors).

Telephone contact by the rehabilitation coach will be organized and the 16-week Stroke Help Cognitive Strategy Training Intervention will proceed. In general the topics or strategies to be discussed will be used to achieve one or more of the following rehabilitation strategies: 1) Understanding cognitive deficits that may result from stroke; 2). Reinforcing, strengthening or re-establishing previously learned patterns of behavior; 3) Establishing new patterns of compensatory mechanisms; 4) Enabling persons to adapt to their cognitive disability.

Following the 16-week Cognitive Strategy Training Intervention participants will have an on-site visit to provide qualitative and quantitative data related to the feasibility and efficacy of the program.

ELIGIBILITY:
Inclusion Criteria:

* history of one or more strokes;
* living in the community;
* subjective concerns about cognitive function;
* ability to give informed consent;
* fluent in written and spoken English.

Exclusion Criteria:

* unstable medical conditions or a co-morbid neurological disorder that could additionally impact cognitive or daily function, such as Parkinson's disease or Multiple Sclerosis;
* no available caregiver or significant other willing to participate in approximately one hour of telephone contact per week with coach and stroke survivor;
* current symptoms of severe depression (Geriatric Depression Scale>20), global aphasia, or dementia (determined by baseline testing).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in functioning on goal attainment scaling | Measured at baseline and week 18
  estimating within subject effect sizes for the treated group based on changes in measures at the level of impairment (self and other-reported cognitive performance), activity (achievement of activity goals and everyday cognitive performance) and participation/quality of life (self-report measures of reintegration to normal living, quality of life, caregiver burden).

SECONDARY OUTCOMES:
Intervention modifiers | measured at baseline and weekly until end of study at week 18
  Additional secondary analyses will also investigate variables that could modify the effects of the interventions, including cognitive profile, stroke severity and location of lesion, co-morbid conditions, type of functional goal and current environmental factors.
Feasibility of recruitment, retention, compliance | measured at end of 16 week study
  Rates of subject recruitment, retention, and compliance with protocol
Feasibility-Coach adherence | measured at weekly intervals
  Feasibility of coach adherence to therapy protocols will be assessed weekly through review of adherence to scripts and completeness of data collection

CONTACTS AND LOCATIONS:
Overall Officials: Gail A Eskes, Ph.D., Principal Investigator — Capital District Health Authority, Nova Scotia, Canada
Locations (1):
- Capital District Health Authority, Halifax, Nova Scotia, Canada